CLINICAL TRIAL: NCT05358288
Title: Investigation of the Effect of Bariatric Surgery on Physical Activity Levels, Spatiotemporal Parameters of Gait, Flexibility and Quality of Life
Brief Title: Effect of Bariatric Surgery on Physical Activity, Gait, Flexibility and Quality of Life
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-235/30
Record Dates: First submitted 2022-04-22; First posted 2022-05-03 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Obesity; Bariatric Surgery; Gait
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to analyze spatio-temporal characteristics of gait, physical activity level and changes in quality of life in patients by measuring conditions before bariatric surgery and third-month after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of obesity
* Body mass index > 35
* Speak and understand Turkish
* Ability of read and write

Exclusion Criteria:

* History of lower extremity surgery
* Musculoskeletal/systemic/neurological/psychiatric problems
* Urinary syndromes
* Limited gait due to cardio-pulmonary insufficiency
* Unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -Having obestity with BMI>35 (indication for bariatric surgery)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
Gait speed | Change from baseline at 3 months
  Participants's gait speed were evaluated by a wearable sensor. This wearable sensor is named BTS G-Walk sensor (BTS Bioengineering S.p.A., Italy) and was attached L4-5 region by a belt. The data were transferred by Bluetooth connection to software while participants' walking.

SECONDARY OUTCOMES:
Support times | Change from baseline at 3 months
  Participants's support times of gait were evaluated by a wearable sensor. The wearable sensor is named BTS G-Walk sensor (BTS Bioengineering S.p.A.,Italy) and was attached L4-5 region by a belt. The data were transferred by Bluetooth connection to software while participants' walking.
Step Length | Change from baseline at 3 months
  Participants's step lengths of gait were evaluated by a wearable sensor. The wearable sensor is named BTS G-Walk sensor (BTS Bioengineering S.p.A.,Italy) and was attached L4-5 region by a belt. The data were transferred by Bluetooth connection to software while participants' walking.
Levels of physical activity | Change from baseline at 3 months
  Physical activity levels were evaluated by the International Physical Activity Questionnaire- Short Form. This form include seven questions. With these questions, it is possible to obtain information about the time individuals spend in walking, moderate and vigorous activities and also time spent sitting. As a result of the calculations, the level of physical activity is divided into three groups. These groups are as follows: Less than 600 metabolic equivalent-minute inactive; between 600-3000 metabolic equivalent-minute are minimum active; more than 3000 metabolic equivalent-minute are very active.
Sit-Reach Test | Change from baseline at 3 months
  The flexibility of the lumbar extensors, hamstrings and gastrocsoleus muscle group was evaluated with the Sit-to-Sit Test. Individuals were asked to sit in a long sitting position, hold their feet in 90 degrees dorsiflexion and reach for their toes with their hands without bending their knees. The test was repeated three times and the mean value was recorded. Positive values were used if this value reached beyond the toes. Higher positive values indicate better flexibility.
Modified Thomas Test | Change from baseline at 3 months
  Flexibility in the Rectus Femoris and Iliopsoas muscles evaluated with "Modified Thomas Test". While bringing her hip to maximum flexion with her hands, she was asked to lower the extremity to be tested towards the ground. Measurements were repeated 3 times for each extremity and these values were average was taken. Measurements were made with a goniometer. Higher values indicate better flexibility.
Popliteal Angle | Change from baseline at 3 months
  Popliteal angle measurement was used for hamstring shortness. The measurement was performed with the participants in supine position with the goniometer zeroed to the anterolateral half of the tibia and the hip stabilized at 90 degrees of flexion. The average of two measurements taken five seconds apart was taken. Values above 20 degrees were considered as hamstring shortness.
Quality of Life | Change from baseline at 3 months
  The Impact of Weight on Quality of Life Questionnaire (IWQOL) was used to assess the participants' quality of life. The scale includes questions on bodily functions, self-esteem, sexual life, social pressure and work. The minimum score that can be obtained from the scale consisting of 31 items in total is 0 and the maximum score is 100. A lower score indicates a lower quality of life.